CLINICAL TRIAL: NCT02117401
Title: A Prospective, Multi-center, Randomized Controlled Study of Neuromuscular Blocking Effect and Safety of Mivacurium Chloride in Pediatric Patients
Brief Title: A Prospective, Multi-center, Randomized Controlled Study of Muscle Relaxation Effect and Safety of Mivacurium Chloride in Pediatric Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20121101
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Efficacy and Safety of Mivacurium Chloride for Pediatric Patients
MeSH Terms: interventions — Mivacurium; Midazolam; Ketamine; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- group 1 (Experimental): age: 2 to 12 months induction dosage of mivacurium chloride: 0.15 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 2 (Experimental): age: 2 to 12 months induction dosage of mivacurium chloride: 0.15 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 3 (Experimental): age: 2 to 12 months induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 4 (Experimental): age: 2 to 12 months induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 5 (Experimental): age: 13 to 35 months induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 6 (Experimental): age: 13 to 35 months induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 7 (Experimental): age: 13 to 35 months induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 8 (Experimental): age: 13 to 35 months induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 9 (Experimental): age: 3 to 6 years induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 10 (Experimental): age: 3 to 6 years induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 11 (Experimental): age: 3 to 6 years induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 12 (Experimental): age: 3 to 6 years induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 13 (Experimental): age: 7 to 14 years induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 14 (Experimental): age: 7 to 14 years induction dosage of mivacurium chloride: 0.20 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 15 (Experimental): age: 7 to 14 years induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 20 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil
- group 16 (Experimental): age: 7 to 14 years induction dosage of mivacurium chloride: 0.25 mg/kg administration: intravenous injection for 40 s
  Interventions: Drug: mivacurium chloride; Drug: midazolam; Drug: ketamine; Drug: propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: mivacurium chloride — intravenously injected during induction with the dose according to allocated group, and intravenously injected with the dose of 0.1 mg/kg when T1 recovers to 25% during period of maintenance.
  Other Names: mivacron
Drug: midazolam — Before induction: after moving into operating room, oral administration with dose of 0.5 mg/kg or mixed with ketamine (midazolam 10 mg+ ketamine 100 mg) with dose of 0.1 ml/kg by intramuscular route for uncooperative children
  Induction: for children who didn't receive mixture of midazolam and ketamine before induction, it will be given with the dose of 0.05 ml/kg
Drug: ketamine — mixed with ketamine (midazolam 10 mg+ ketamine 100 mg) with dose of 0.1 ml/kg by intramuscular route for uncooperative children
  Induction: for children who didn't receive mixture of midazolam and ketamine before induction, it will be given with the dose of 0.05 ml/kg
Drug: propofol — Induction: 2 to 3 mg/kg Maintenance: 50 to 100 mcg/kg/min
Drug: Remifentanil — Induction: 2 mcg/kg Maintenance: 0.1 to 0.3 mcg/kg/min

SUMMARY:
To evaluate the effect and safety of mivacurium chloride in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* The parent/guardian must sign a parental permission consent document
* American Society of Anesthesiologists (ASA) physical status class 1-3
* Elective surgery patients with tracheal intubation, and the operation duration is expected to be longer than 30 min but no longer than 120 min(cleft lip and palate, orthopedic, bilateral hernia, bilateral cryptorchidism, hypospadias crack, and other ear, nose and throat surgery, etc)
* Age between 2 months to 14 Years

Exclusion Criteria:

* BMI<18kg/m2 or BMI>31kg/m2
* Patients with serious respiratory, cardiovascular disease, and liver and kidney dysfunction[AST（glutamic oxalacetic transaminase）,ALT(glutamic-pyruvic transaminase)>1.5 Normal;BUN(blood urea nitrogen)>Normal)]
* Patients with asthma or airway hyperresponsiveness, neuromuscular patients disease or cachexia
* Preoperative hemoglobin less than 10g/L
* Hypoproteinemia TP（total protein) <45g/L
* Diabetic patients
* Patients with difficulty airway
* Patients with Known or suspected atypical plasma cholinesterase gene homozygous
* Burn patients
* Patients with serious acid-base imbalances, or severe electrolyte imbalance
* Patients with neuromuscular relaxants in a week
* Patients prohibited with muscle relaxants, or allergy to any component of mivacurium
* Patients participated in any drug clinical trial with 30 days before the start of the study
* Other situations not suitable for inclusion
* Blood loss more than 10 ml/kg in surgery

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1152 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
intubation score | 1 minute within intubation
  Krieg Tracheal Intubation Score
  * Score ： 1 2 3 4
  * Laryngoscopy ： Easy Fair Difficult Impossible
  * Vocal cords： Open Moving Closing Closed
  * Coughing： None Diaphragm Mild Severe
  * A total score of 3-4 = excellent, 5-7 = good, 8-10 = poor, 11-12 = bad.
muscle relaxation effect | from baseline to no more than 120 minutes after intubation
  * Recording T1 and TOFR（Train of four ratio) before/after the induction of anesthesia -Onset time of Mivacurium：time from end of injection until occurrence of maxi- mum block
  * Duration of clinical relaxation：time to recovery of Tl(the first response in the TOF) to 25%
  * Recovery index：Time interval during with T1 recovered from 25%

REFERENCES:
- [Derived] Zeng R, Liu X, Zhang J, Yin N, Fei J, Zhong S, Hu Z, Hu M, Zhang M, Li B, Li J, Lian Q, ShangGuan W. The efficacy and safety of mivacurium in pediatric patients. BMC Anesthesiol. 2017 Apr 17;17(1):58. doi: 10.1186/s12871-017-0350-2. PMID 28415988